CLINICAL TRIAL: NCT04549987
Title: Speed of Premolar Extraction Space Closure: The Effect of Every Visit Replacement of Working Arch Wire - A Prospective Randomized Clinical Trial
Brief Title: Speed of Premolar Extraction Space Closure: Every Visit Replacement of Working Archwire
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Elham Abu Alhaija, Professor, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 53/2019
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Orthodontic Appliance
Keywords: Tooth movement; Friction; Rate

STUDY DESIGN:
Intervention Model Description: Working archwire status
Who Masked: Participant, Outcomes Assessor
Masking Description: The intervention was randomly allocated to either the right or left side using the permuted random block size of 2 with 1:1 allocation ratio. The random sequences for each intervention to either right or left sides was concealed in opaque envelopes and shuffled before the intervention to increase the unpredictability of the random allocation sequence. Each patient was asked to pick a sealed envelope to assign the intervention to either the right or left side. Allocation concealment was aimed to prevent selection bias and to protect the assignment sequence until allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Without changing working archwire (Experimental): Extraction space closed using the same working archwire throughout 3 visits after insertion
  Interventions: Device: Space closure without changing working archwire monthly
- With changing working archwire (Experimental): The extraction space closed having the working archwire changed monthly.
  Interventions: Device: Space closure withchanging working archwire monthly

INTERVENTIONS:
Device: Space closure without changing working archwire monthly — Upper premolar space closure using the same 0.019X0.025 stainless steel archwire every month
  Arms: Without changing working archwire
Device: Space closure withchanging working archwire monthly — Upper premolar space closure using new 0.019X0.025 stainless steel archwire every month
  Arms: With changing working archwire

SUMMARY:
The aims of this trial were to assess the effect of changing 0.019X0.025-inch SS working archwire monthly on the rate of space closure, to compare the frictional resistance of unchanged and new working archwires in-vitro, and to assess its effect on the rate of space closure, to record the amount of ion concentration in the saliva before orthodontic treatment, before space closure and one month after space closure.

DETAILED DESCRIPTION:
The aims were to assess the effect of changing 0.019X0.025-inch SS working archwire monthly on the rate of space closure, to compare the frictional resistance of unchanged and new working archwires in-vitro and to assess its effect on rate of space closure, to record the amount of ion concentration in the saliva before orthodontic treatment, before space closure and one month after space closure and to compare the rate of teeth movement into fresh and old extraction sites.

Trial design: Randomized controlled clinical trial with a split-mouth design. Setting: Jordan University of Science and Technology(JUST) Postgraduate Dental Teaching Clinics and labs.

Participants and interventions: Twenty-eight subjects with bimaxillary proclination requiring extraction of all first premolar teeth participated in this study. In the upper arch two groups were identified; group 1 having the extraction space closed using the same working archwire throughout 3 visits after insertion, and group 2 with the working archwire changed monthly.

The working archwire in the upper arch was split into 2 halves in the midline and each one half was connected to the other by a wide joining hook. Patients were followed-up monthly for three months. At every follow up visit upper alginate impressions were taken and the working archwire in the upper arch was changed on one side only. Upper follow-up models were scanned using digital scanner and spaces were measured using digital software.

Three unstimulated saliva samples were collected from each patient; prior to commencement of treatment, when 0.019X0.25-inch SS archwire was reached and before space closure and one month after space closure.

The rate of extraction space closure in the upper arch, ion concentration in saliva samples measured using inductively coupled plasma mass spectrometer (ICP-MS) and frictional resistance of the working archwires was measured using universal mechanical testing machine.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 16 years
* Proclined upper and lower incisors (Ui/max >115 o, Li/mand >99o)
* Mild upper and lower arch crowding (<4mm) or no crowding
* Need for upper and lower first premolars extraction
* Skeletal I malocclusion (1<ANB <5)
* Average lower facial height and maxillomandibular plane angle (22 o <MM<32 o)
* Class I canine relationship
* Good oral hygiene and healthy periodontium

Exclusion Criteria:

* Poor oral hygiene
* Diseases and medications that were likely to affect bone biology
* Previous orthodontic treatment
* Evidence of bone loss
* Active periodontal disease
* Smoking

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
The amount of space closure per month | 3 months
  the width of upper extraction space in milimeters

SECONDARY OUTCOMES:
ion concentration in saliva | through study completion, an average of 1 year
  Concentration of ions (Chrome, Iron, Nickel, titanium) in saliva
Frictional resistance | At the end of the study
  A mean value in N for frictional force over a 3 millimeter distance.

CONTACTS AND LOCATIONS:
Overall Officials: Elham S A Alhaija, PhD, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Faculty of Dentistry/Jordan University of Science and Technology Dental Teaching Clinics, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No